CLINICAL TRIAL: NCT05385809
Title: A Retrospective Study of Sintilimab Combined With Chemotherapy in Conversion Therapy of Unresectable Locally Advanced or Stage IV Gastric Cancer/Gastroesophageal Junction Carcinoma
Brief Title: A Retrospective Study of Immunotherapy in Conversion Therapy of Unresectable Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Innovent Biologics, Inc. (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, MD, Zhejiang Cancer Hospital
Other Study IDs: IRB-2022-278
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Unresectable Gastric Cancer
Keywords: Unresectable Gastric Cancer; Conversion Therapy; Immunotherapy; Sintilimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was an observational, non-interventional, multicenter retrospective study to evaluate the feasibility and safety of sintilimab combined with chemotherapy (SOX or PS) in the clinical practice of unresectable locally advanced or stage IV gastric cancer/gastroesophageal junction carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18-75 Years (concluding 18 and 75 Years)
* Pathologically confirmed gastric/gastroesophageal junction adenocarcinoma
* Unresectable, locally advanced or limited distant metastasis of IV gastric cancer(AJCC 8th)
* Meets only ≤2 of the following conditions: highly locally advanced (T4b), or extensive or bulcky lymph nodes; Para-aortic lymph node metastasis(mainly 16A2/B1 region); limited liver metastasis(H1); limited Peritoneal metastasis(CY1, P1), with or without ovarian metastasis(Kukernburg tumor);
* Untreated(e.g. radiotherapy, chemotherapy, target therapy, immunotherapy, et al.)
* At least 1 measurable lesion by RECIST v1.1 criteria
* ECOG PS: 0-2
* Received sintilimab combined with chemotherapy(SOX or PS) at least 1 cycle

Exclusion Criteria:

* Known Her2 positive
* Patients with incomplete data or other factors affecting the judgment of efficacy and safety

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 pantients with histologically confirmed GC/esophagogastric junction cancer (EGJC) who received immunotherapy prior to surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical conversion rate | two years

SECONDARY OUTCOMES:
R0 resection rate | two years
  Defined as no residue under the microscope after resection
Major pathological response (MPR) | two years
  MPR is defined as less than 10% residual tumor after neoadjuvant therapy
Overall response rate ( ORR) | two years
  ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR or PR according to RECIST 1.1 based on investigator assessment
adverse event (AEs) | two years

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, MD, PhD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China